CLINICAL TRIAL: NCT06171022
Title: The Effect of Cherry Seed Pillow on Pain and Quality of Life in Patients With Fibromyalgia
Brief Title: The Effect of Cherry Seed Pillow on Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Gerçek (Other)
Responsible Party: Sponsor-Investigator, Hasan Gerçek, Lecturer, KTO Karatay University
Organization: KTO Karatay University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KaratatUH10
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cherry seed pillow (Experimental): 4 Weeks, 5 days a week, 20 minutes, in addition to the physiotherapy application of the routine, a heated cherry seed pillow will be applied.
  Interventions: Other: Cherry seed pillow
- Control (Active Comparator): 4 Weeks, 5 days a week, 20 minutes, in addition to the physiotherapy application of the routine, a hot-pack will be applied.
  Interventions: Other: Control

INTERVENTIONS:
Other: Cherry seed pillow — 4 Weeks, 5 days a week, in addition to the routine physiotherapy application, 20 minutes of heated cherry seed pillow will be applied to the participant's back area.
  Arms: Cherry seed pillow
Other: Control — 4 Weeks, 5 days a week, in addition to the routine physiotherapy application, 20 minutes of hotpack will be applied to the participant's back area.
  Arms: Control

SUMMARY:
In this study, the effects of 4-week Cherry seed pillow application on pain and quality of life in individuals diagnosed with fibromyalgia will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Diagnosis of Fibromyalgia according to ACR classification criteria
* Neuromuscular system examination is normal
* Pain (vas-visual anologous scale) level of at least 5 points
* No communication problems
* Willingness to participate in the practice of using cherry seed cushion
* To be capable of answering the data collection tools to be used in the research
* Not having made hot, cold etc. applications at home

Exclusion Criteria:

* -No diagnosis of Fibromyalgia according to ACR classification criteria
* Normal examination of the neuromuscular system
* Pain (vas-visual anologous scale) level between 0-5
* Communication problems
* Failure to accept the practice of using cherry seed cushion and failure to finish the implementation process
* Having a musculoskeletal disorder other than fibromyalgia
* Pregnant or lactating
* To be capable of answering the data collection tools to be used in the research
* Having made hot, cold etc. applications at home

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain at 4 weeks | Baseline and 4 weeks
  he rest, activity and night pains of the participants will be evaluated with a 10 cm Visual Analog Scale before the treatment and at the end of the 4-week application. "0" means no pain, "10" means excruciating pain. Results will be recorded in cm.

SECONDARY OUTCOMES:
Change from baseline in function at 4 weeks | Baseline and 4 weeks
  The Fibromyalgia Impact Questionnaire will be used to assess the functioning of the participants. The questionnaire consists of 20 questions. As the score increases, the function decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)